CLINICAL TRIAL: NCT05841771
Title: A Single Arm, Phase 2 Study Evaluating Safety and Efficacy of Maintenance Therapy With Hypomethylating Agent and Venetoclax After Allogeneic Stem Cell Transplantation in Patients With f High-risk Myeloid Malignancies.
Brief Title: Hypomethylating Agent and Venetoclax After Allo-HSCT in Patients With High-risk Myeloid Malignancies.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liping Wan, Associate Director of Department of Hematology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-AZA-VEN-202301
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hypomethylating Agent; Venetoclax; Myeloid Malignancy
MeSH Terms: interventions — venetoclax; PTH2 protein, human; Azacitidine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZA-VEN maintenance (Experimental): hypomethylating agents (azacytidine 32mg/m2 or decitabine 5mg/m2) for 5 days and venetoclax 400mg/d for 7 days, repeated every 28 days until up to 1-year posttransplant.
  Interventions: Drug: Venetoclax; Drug: Azacitidine or decitabine

INTERVENTIONS:
Drug: Venetoclax — Participants will receive maintenance therapy with venetoclax and azacitidine or decitabine after allogeneic stem cell transplantation.
  Azacitidine will be administered once daily subcutaneously (32mg/m2/d) on days 1-5, and venetoclax will be administered once daily orally (400mg/day) on days 1-7. If the patient is refractory or allergic to azacitidine, they will receive decitabine. Decitabine will be administered intravenously (5mg/m2/d) on days 1-5. If the patient is treated with CYP450 inhibitors(such as posaconazole or voriconazole), the dose of venetoclax will reduce to 100 mg once daily on days 1-7. Maintenance therapy will start from the 60th to 120th days after allogeneic hematopoietic stem cell transplantation and repeat every 28 days for up to 10 cycles within the first year after transplantation.
  Other Names: BCL-2 inhibitor
Drug: Azacitidine or decitabine — azacytidine 32mg/m2 or decitabine 5mg/m2
  Other Names: Hypomethylating Agent

SUMMARY:
The main objective of the study is to evaluate the efficacy and safety of maintenance therapy with hypomethylating agent and Venetoclax to improve leukemia free survival for high-risk myeloid malignancies after allogeneic hematopoietic stem cell transplantation .

DETAILED DESCRIPTION:
This is a prospective single-arm study. Patients with high-risk AML or MDS aged between 18-70 years old will enroll in the study. They will be given hypomethylating agents (azacytidine 32mg/m2 or decitabine 5mg/m2) for 5 days and venetoclax 400mg/d for 7 days after allogeneic hematopoietic stem cell transplantation. The maintenance therapy will start from 60th days posttransplant, repeated every 28 days until up to 1-year posttransplant. The 1-year leukemia-free survival rate，1-year cumulative recurrence rate, and 1-year overall survival will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML or MDS and have received allogeneic hematopoietic cell transplantation;
* Patients with AML must have one of the following high-risk factors: Cytogenetics and molecular features consistent with adverse risk group by European LeukemiaNet classification for AML； require more than 2 courses of induction chemotherapy to reach complete remission； Extramedullary myeloid malignancy；≥CR2； Presence of measurable residual disease at the time of HSCT. *
* Patients with MDS must have one of the following high-risk factors: IPSS-R scores are high-risk or very high-risk； Presence of TP53 mutation； Presence of measurable residual disease at the time of HSCT. *
* CBC: ANC ≥ 1.0 × 10e9/L, Hb ≥ 80g/L, and PLT ≥ 50 × 10e9/L；
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

  * Presence of measurable residual disease at the time of HSCT is defined as the following: Blast percentage in bone marrow detected by flow cytometry ≥0.01%； Presence of fusion gene or mutated gene by qPCR.

Exclusion Criteria:

* Concurrent use of targeted drugs ;
* Resistant to Venetoclax before transplantation;
* Allergic to decitabine , Azacitidine or venetoclax;
* Active grade II or higher acute GVHD ;
* Active moderate or severe chronic GVHD ;
* Diseases recurrence (abnormal myeloid cells detected by flow cytometry >0.01%, presence of WT1 or other genes, or extramedullary malignancy ), percentage of donor cells in bone marrow <90% or graft rejection:
* CBC: ANC < 1.0 × 10e9/L, or PLT < 50 × 10e9/L；
* Severe organ dysfunction: Elevated Aspartate transaminase (AST) /alanine transaminase (ALT), or direct bilirubin >3 times upper limit of normal; Creatinine clearance (Ccr)<50mL/min or serum creatinine >1.5 times upper limit of normal, whether hemodialysis treatment is performed;
* Active uncontrolled systemic fungal, bacterial, or viral infection
* Pregnant or lactating women;
* Other severe complications and not suitable judged by researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Leukemia-free survival (LFS) time | From the date of transplantation, assessed up to 1 year after transplantation.
  Summary statistics for LFS time will be computed for all patients.

SECONDARY OUTCOMES:
Cumulative incidence of relapse | From the date of transplantation, assessed up to 1 year after transplantation.
  Use the method of Gooley et al to estimate the cumulative incidence of relapse.
Overall survival | From the date of transplantation, assessed up to 1 year after transplantation.
  The method of Kaplan and Meier will be used to estimate the distribution of overall survival. Cox proportional hazards regression analysis will be used to model the association between overall survival and covariates of interest.
Incidence of toxicity of the regimen | From the date of transplantation, assessed up to 1 year after transplantation.
  Descriptive statistics will be used to summarize adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Liping Wan, M.D., Principal Investigator — Shanghai Jiao Tong University School of Medicine Affiliated Shanghai General Hospital
Locations (1):
- Shanghai Jiao Tong University School of Medicine Affilated Shanghai General Hospital, Shanghai, Shanghai Municipality, China